CLINICAL TRIAL: NCT01194843
Title: A Double-blind Placebo-controlled Evaluation of Ropivacaine Efficacy by Local Per and Post Hepatectomy Infiltrations for Adult Pain Management
Brief Title: Placebo-controlled Evaluation of Ropivacaine Efficacy by Local Infiltrations
Acronym: DPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: AstraZeneca (Industry); Fondation Apicil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: DPO-Hepatectomy; ET2007-073 (Registry Identifier: Centre Léon Bérard); 2007-007968-19 (EudraCT Number)
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2014-01

CONDITIONS: Hepatectomy; Pain; Metastasis
MeSH Terms: conditions — Pain; Neoplasm Metastasis | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine (Experimental): Ropivacaine administration by local per and post surgery infiltration
  Interventions: Drug: Ropivacaine
- Physiological serum (Active Comparator): Administration of physiological serum by local per and post surgery infiltration
  Interventions: Drug: Physiological serum

INTERVENTIONS:
Drug: Ropivacaine — 40 ml infiltration at the end of the hepatectomy and then continuous local infiltration of 8 ml per hour over the 4 days after the hepatectomy
  Arms: Ropivacaine
Drug: Physiological serum — 40 ml infiltration at the end of the hepatectomy and then continuous local infiltration of 8 ml per hour over the 4 days after the hepatectomy
  Arms: Physiological serum

SUMMARY:
The purpose of the study is to evaluate the efficacy and impact on morphine consumption of ropivacaine administered by local per and post hepatic surgery infiltration.

Patients will be randomized to either ropivacaine or physiological serum, with equivalent administration modalities in both arms.

Patients will be followed during 4 days after the surgery. They will also come back for a follow-up visit one month later.

It is necessary to enrol 100 patients. The estimated period of inclusion is 24 months.

This is a prospective, comparative, monocentric, double-blind randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18 years
* Patients with histologically confirmed cancer
* Patients treated at the Centre Léon Bérard
* Patients requiring a surgery for hepatic metastases
* ASA <= 3
* At least 3 weeks between surgery and chemotherapy
* Total bilirubin < 1.5 x upper limit of normal range
* ASAT and ALAT < 5 times x upper limit of normal range
* Creatinine clearance > 60 ml per hour
* Serum creatinine < 115 µmol/l
* Mandatory affiliation with a health insurance system
* Patients able to understand French
* Signed, written informed consent

Exclusion Criteria:

* Patients with a hepatocellular carcinoma or an initial liver cancer
* Patients treated chronically by morphine
* Patients that already have abdominal pain
* Patients who are allergic either to morphinics, local anesthesics, paracetamol, NSAID or cortisone
* Patients suffering from heart, kidney or liver insufficiency
* Documented history of cognitive or psychiatric disorders
* Pregnant or lactating women
* Difficult follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2009-03; Primary Completion 2014-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of ropivacaine versus physiological serum administered by local infiltration and impact on morphine consumption | In the 4 days following the hepatectomy

SECONDARY OUTCOMES:
Efficacy of ropivacaine versus physiological serum administered by local infiltration and impact on daily morphine consumption | In the 4 days following the hepatectomy
Evaluation of patients' perception of post-surgery pain | In the 4 days following the hepatectomy
Immediate and late complications related to the perfusion, the medical device and other predictable side effects | In the 4 days following the hepatectomy and one month later
Patients' post-surgery rehabilitation | Between surgery and follow-up visit, one month later
Patients' satisfaction with the pain care | Four days after the hepatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Peres-Bachelot, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard, Lyon, France

REFERENCES:
- [Background] Beaussier M, El'Ayoubi H, Schiffer E, Rollin M, Parc Y, Mazoit JX, Azizi L, Gervaz P, Rohr S, Biermann C, Lienhart A, Eledjam JJ. Continuous preperitoneal infusion of ropivacaine provides effective analgesia and accelerates recovery after colorectal surgery: a randomized, double-blind, placebo-controlled study. Anesthesiology. 2007 Sep;107(3):461-8. doi: 10.1097/01.anes.0000278903.91986.19. PMID 17721249
- [Background] Bianconi M, Ferraro L, Ricci R, Zanoli G, Antonelli T, Giulia B, Guberti A, Massari L. The pharmacokinetics and efficacy of ropivacaine continuous wound instillation after spine fusion surgery. Anesth Analg. 2004 Jan;98(1):166-172. doi: 10.1213/01.ANE.0000093310.47375.44. PMID 14693613
- [Background] Borromeo CJ, Stix MS, Lally A, Pomfret EA. Epidural catheter and increased prothrombin time after right lobe hepatectomy for living donor transplantation. Anesth Analg. 2000 Nov;91(5):1139-41. doi: 10.1097/00000539-200011000-00018. PMID 11049898
- [Background] Godier A, Babinet A, el Metaoua S, Fulgencio JP, Bonnet F. [A new cause of postoperative confusion syndrome: nefopam]. Ann Fr Anesth Reanim. 2002 Jun;21(6):538-9. doi: 10.1016/s0750-7658(02)00650-0. French. PMID 12134601
- [Background] Ho AM, Lee A, Karmakar MK, Samy W, Lai PB, Ho OA, Cho A. Hemostatic parameters after hepatectomy for cancer. Hepatogastroenterology. 2007 Jul-Aug;54(77):1494-8. PMID 17708283
- [Background] Jalan R, Williams R, Bernuau J. Paracetamol: are therapeutic doses entirely safe? Lancet. 2006 Dec 23;368(9554):2195-6. doi: 10.1016/S0140-6736(06)69874-7. No abstract available. PMID 17189017
- [Background] Kwan AL. Epidural analgesia for patient undergoing hepatectomy. Anaesth Intensive Care. 2003 Apr;31(2):236-7. No abstract available. PMID 12712800
- [Background] Larson AM. Acetaminophen hepatotoxicity. Clin Liver Dis. 2007 Aug;11(3):525-48, vi. doi: 10.1016/j.cld.2007.06.006. PMID 17723918
- [Background] Liu SS, Richman JM, Thirlby RC, Wu CL. Efficacy of continuous wound catheters delivering local anesthetic for postoperative analgesia: a quantitative and qualitative systematic review of randomized controlled trials. J Am Coll Surg. 2006 Dec;203(6):914-32. doi: 10.1016/j.jamcollsurg.2006.08.007. Epub 2006 Oct 25. No abstract available. PMID 17116561
- [Background] Mazoit JX, Butscher K, Samii K. Morphine in postoperative patients: pharmacokinetics and pharmacodynamics of metabolites. Anesth Analg. 2007 Jul;105(1):70-8. doi: 10.1213/01.ane.0000265557.73688.32. PMID 17578959
- [Background] Murphy EJ. Acute pain management pharmacology for the patient with concurrent renal or hepatic disease. Anaesth Intensive Care. 2005 Jun;33(3):311-22. doi: 10.1177/0310057X0503300306. PMID 15973913
- [Background] Schumann R, Zabala L, Angelis M, Bonney I, Tighiouart H, Carr DB. Altered hematologic profiles following donor right hepatectomy and implications for perioperative analgesic management. Liver Transpl. 2004 Mar;10(3):363-8. doi: 10.1002/lt.20059. PMID 15004762
- [Background] Tsui SL, Yong BH, Ng KF, Yuen TS, Li CC, Chui KY. Delayed epidural catheter removal: the impact of postoperative coagulopathy. Anaesth Intensive Care. 2004 Oct;32(5):630-6. doi: 10.1177/0310057X0403200503. PMID 15535484
- [Background] Urwin SC, Smith HS. Fatal nefopam overdose. Br J Anaesth. 1999 Sep;83(3):501-2. doi: 10.1093/bja/83.3.501. PMID 10655934
- [Background] Villier C, Mallaret MP. Nefopam abuse. Ann Pharmacother. 2002 Oct;36(10):1564-6. doi: 10.1345/aph.1C017. PMID 12243607
- [Background] Ychou M, Viret F, Kramar A, Desseigne F, Mitry E, Guimbaud R, Delpero JR, Rivoire M, Quenet F, Portier G, Nordlinger B. Tritherapy with fluorouracil/leucovorin, irinotecan and oxaliplatin (FOLFIRINOX): a phase II study in colorectal cancer patients with non-resectable liver metastases. Cancer Chemother Pharmacol. 2008 Jul;62(2):195-201. doi: 10.1007/s00280-007-0588-3. Epub 2007 Sep 28. PMID 17901955